CLINICAL TRIAL: NCT04894539
Title: Transcutaneous Electrical Nerve Stimulation as a Pain-relieving Approach in Labor Pain Control: a Randomized Double-blinded Controlled Pilot Study
Brief Title: Transcutaneous Electrical Nerve Stimulation for Labor Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Centaflow (Industry); Herning Hospital (Other)
Responsible Party: Principal Investigator, Kenoja Thuvarakan, Principle Investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20190821
Record Dates: First submitted 2021-05-13; First posted 2021-05-20 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Labor Pain
Keywords: TENS; Labor pain; Childbirth; RCT; Pilot study
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: 3 groups (TENS1, TENS2, and sham)
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TENS1 (Experimental): TENS with 4/100 Hz in frequency, 200 µs in pulse duration, and intensity individually adjusted.
  Interventions: Device: DS5 electrical stimulator
- TENS2 (Experimental): TENS with 80/100 Hz in frequency, 200 µs in pulse duration, and intensity individually adjusted.
  Interventions: Device: DS5 electrical stimulator
- Sham-TENS (Sham Comparator): Sham with 100 Hz in frequency, 200 µs in pulse duration, and intensity below 5 mA.
  Interventions: Device: DS5 electrical stimulator

INTERVENTIONS:
Device: DS5 electrical stimulator — TENS

SUMMARY:
Transcutaneous electrical nerve stimulation (TENS) is a non-invasive electro-physical modality used for several pain conditions including labor pain control. Despite several years of research, there is still no agreement within the literature regarding the selection of TENS parameters. It is aimed to investigate two types of TENS frequencies (TENS1 alternating between 4 to 100 Hz and TENS2 alternating between 80 to 100 Hz) compared to sham-TENS.

DETAILED DESCRIPTION:
Midwives and the study investigator will ask parturients, who are admitted to the labor ward at Region Hospital Herning satisfying the inclusion and exclusion criteria, whether they are interested in attending the experimental session.

The study will be conducted as soon as the subject is admitted at the labor ward. The study will only be conducted during early and active labor and not during the birth of the baby.

The subject in this study includes the package of a parturient and her neonate (after birth) as we also obtain data about the neonate. Hereby, two consent forms will be obtained. As this study is a non-invasive study, it is decided to have at least the consent of one parent.

The investigator will fill out a questionnaire about the parturient in cooperation with the subject and midwife, including screening questions related to inclusion and exclusion criteria before the experimental session starts.

The study will last approximately one hour and will be conducted during laboring circumstances. KT (Kenoja Thuvarakan) will carry out the experiment, and she will be present in the delivery room during the whole session.

The study includes several outcomes, including subjective and semi-objective pain measures. The primary outcome is VAS (0-10 cm scale), while secondary outcomes include PPT and satisfaction questionnaire (only at the end of the study). The subjects will be asked before, and immediately after the experimental exposure about the four outcomes (VAS and PPT). The subjects will be exposed to one of the two combinations of TENS stimulation (low and high alternating frequency), which will be compared to sham-TENS.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Between ages 18-39 years
* Vertex presentation
* Speak, read and understand Danish
* At term (37-42 weeks gestation age)

Exclusion Criteria:

* High-risk pregnancies (including risk factors: eclampsia, pre-eclampsia, diabetes, gestational diabetes, hypertension, and hypotension, intrauterine growth restriction, polyhydramnios, and oligohydramnios).
* Pre-gestational body mass index above 40 kg/m2
* Use of fetal-scalp electrode during the experiment
* Use of pacemakers and other electronic implants
* Severe arrhythmia
* Present musculoskeletal/neurological illnesses
* Chronic pain within last 6 months
* Present medicated mental disorders
* Dermatological disorders
* Use of other long-acting pain relief
* Use of TENS 48 hours before the trial
* Drug addiction defines as the use of cannabis, opioids, or other drugs.
* Smokers
* Lack of ability to cooperate

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog scale (VAS) | Baseline, 10 minutes post stimulation, 30 minutes post stimulation
  10-cm pain intensity scale with 0 cm is no pain and 10 cm is unbearable pain. Decreased cm after baseline measurement indicates pain relief.
Change in Pain pressure threshold | Baseline, 10 minutes post stimulation, 30 minutes post stimulation
  Pain sensitivity measurement also defined as the minimum pressure needed to evoke a pain response measured in kPa. Increased kPa after baseline measurement indicates pain relief.

SECONDARY OUTCOMES:
Satisfaction of TENS | Right after last measurements of VAS & PPT
  Satisfaction rating on scale from 0 to 10 [0 as 'no satisfaction' and 10 as 'total satisfaction'].
Experienced pain reduction | Right after last measurements of VAS & PPT
  Response to yes or no
Interest in the use of TENS again | Right after last measurements of VAS & PPT
  Response to yes, no, or don't know
Recommend TENS to others | Right after last measurements of VAS & PPT
  Response to yes, no, or don't know

CONTACTS AND LOCATIONS:
Overall Officials: Parisa Gazerani, PhD, Study Director — Aalborg University
Locations (1):
- Region Hospital Gødstrup, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data is described in Danish and therefore no plan of sharing.